CLINICAL TRIAL: NCT05918562
Title: Efficacy of a Low Fiber Diet for Pediatric Colonoscopy Prep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Michael Herzlinger, MD, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1640783-12
Record Dates: First submitted 2023-05-31; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Colitis; Gastrointestinal Diseases; Pediatric Disorder; Pediatric Crohns Disease; Procedural Sequelae
MeSH Terms: conditions — Colitis; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low fiber diet group (Experimental): Subjects are allowed a low fiber diet the day of their colonoscopy prep
  Interventions: Dietary Supplement: Low fiber diet
- Clear liquid diet group (Active Comparator): Subjects are allowed a clear liquid diet the day of their colonoscopy prep, as is standard of care
  Interventions: Dietary Supplement: Standard clear liquid diet

INTERVENTIONS:
Dietary Supplement: Low fiber diet — Low fiber diet including cereal, white bread, eggs, meat, dairy
  Other Names: Experimental group
  Arms: Low fiber diet group
Dietary Supplement: Standard clear liquid diet — Standard clear liquid diet including broth, jello, water, juice
  Other Names: Standard group
  Arms: Clear liquid diet group

SUMMARY:
This study is designed to evaluate if pediatric patients who are undergoing a bowel preparation in anticipation of a colonoscopy may be able to take in a low fiber diet instead of a standard, clear liquid diet, while still accomplishing an adequate bowel prep.

ELIGIBILITY:
Inclusion Criteria:

- All outpatients undergoing colonoscopy at our institution

Exclusion Criteria:

* Unstable medical condition
* Metabolic disease
* Inpatient status
* Requiring an emergency colonoscopy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Prep Score | immediately after the colonoscopy
  Scale from 0 - 3 (0 = Unprepared segment colon; 3 = well-visualized segment of colon)

SECONDARY OUTCOMES:
Patient tolerance | immediately before the colonoscopy
  Internally developed questionnaire inquiring patients about their experience with their prep including likert scale measures of hunger, fullness, nausea, stress, and ease of compliance to regimen)

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No